CLINICAL TRIAL: NCT00521677
Title: Comparison Between Two Methods of Oral Care on the Incidence of VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAP1
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: VAP; Oral care; Acquired pneumonia; Mortality; LOS in ICU; LOS in hospital; All patients on ventilator in the ICU
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Procedure: Use of protocol that use special suction connected toothbrush to clean the teeth and the oral cavity, use of non alcoholic antiseptic solution and lubrication of the lips and the oral cavity.
  Interventions: Procedure: Sage oral care
- 2 (Active Comparator): The traditional method of oral care with cleaning of the oral cavity with a sponge soaked with antiseptic non alcoholic solution
  Interventions: Procedure: Traditional oral care

INTERVENTIONS:
Procedure: Sage oral care — Oral care include teeth brush and oral cavity cleaning with a non alcoholic solution, TID
  Arms: 1
Procedure: Traditional oral care — Cleaning of oral cavity with menthol solution, TID
  Other Names: Tarodent
  Arms: 2

SUMMARY:
Patients on ventilator are in high risk to develop ventilator associated pneumonia (VAP). This acquired infection significantly increases morbidity and mortality of these patients.

Studies that investigated the factors influencing the incidence of VAP proved that infectious agents located in the throat and oral cavity are important factors.

The assimilation of oral cavity treatment, including teeth brushing, cleaning and removal of secretions may significantly decrease the incidence of VAP. Choosing the method of oral cavity cleaning is based on few studies that demonstrated the optimal influence of combining mechanical cleansing, the use of a non alcoholic antiseptic material and lubrication of the lips and the oral cavity. Most of these studies are retrospective. The study will compare the traditional method of oral cavity treatment with the use of protocol that use special suction connected toothbrush to clean the teeth and the oral cavity, use of non alcoholic antiseptic solution and lubrication of the lips and the oral cavity.

The current study is a prospective, open label, statistically balanced study that will investigate the connection between the method of oral cavity treatment and the incidence of VAP. 100 patients will be included.

All ventilated patients in the ICU will be eligible and will be included after an informed consent will be signed by the patient, or by his legal guardian. Exclusion criteria include age less than 18 y/o, pregnancy, expected survival of less than 48 hours, immunosupression (excluding patients on steroids), severe burns, existing pneumonia and patient already included in another study.

The main outcome will be 30 days all cause mortality. Secondary outcomes include the development of VAP, days on ventilator, LOS in the ICU and LOS in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* All ventilated patients in the ICU
* Older than 18 y/o

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Immunosuperessed patients
* Expected survival of less than 48 hours
* Burns
* Existing pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The influence of oral care, including teeth brush and oral cavity cleaning with non alcoholic solution in ventilated ICU patients, on the incidence of VAP | 30 days

SECONDARY OUTCOMES:
30 days all cause mortality, days off ventilator, LOS in ICU, LOS in hospital, use of antibiotics | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Amiram Lev, MD, Principal Investigator — HaEmek MC; Tzipi Yakoby, RN, MA, Study Director — HaEmek MC
Locations (1):
- General Intensive Care Unit, HaEmek MC, Afula, Israel